CLINICAL TRIAL: NCT05911191
Title: Can Resistance Training Bring Additional Benefits to a Cardiac Surgery Exercises Based Prehabilitation Program? Protocol for a Non-randomized Controlled Clinical Study of Valvular Heart Disease Patients. Cardiac EBPrehab.
Brief Title: Preoperative Strength-resistance Training in Valvular Heart Disease Patients
Acronym: CardiacEBPhb
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cardenal Herrera University (Other)
Collaborators: Hospital de la Ribera (Other); University of Valencia (Other)
Responsible Party: Principal Investigator, JORGE MONTERO CÁMARA, PhD Student, Cardenal Herrera University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PI 04-05/23
Record Dates: First submitted 2023-06-12; First posted 2023-06-20 (Actual); Last update posted 2023-06-20 (Actual); Status verified 2023-06

CONDITIONS: Exercise Based Prehabilitation in Valvular Surgery
Keywords: Physiotherapy; Muscular strengthening; Quality of life; Hospital stay

STUDY DESIGN:
Intervention Model Description: A prospective, parallel, non-randomised, single-centre, clinical trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: None of the evaluators or caregivers will know the group assignment of each participant. The person responsible for analyzing the data will only see on the data sheet whether they belong to group 1 or group 0, but they will not know which group each of the values is assigned to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Both groups will receive a first session in which they will be instructed to carry out the unsupervised home EBPrehab program, consisting of respiratory training, ventilatory training, strengthening of the respiratory muscles, aerobic endurance exercise through continuous walking, and a series of recommendationss on post-surgical care
- Experimental (Experimental): Addittionally, a preoperative musculoskeletal and cardiopulmonary rehabilitation program focused on peripheral resistance training, will be implemented in the experimental group
  Interventions: Other: Exercise based prehabilitation

INTERVENTIONS:
Other: Exercise based prehabilitation — A peripheral muscle strengthening program
  Arms: Experimental

SUMMARY:
Cardiovascular diseases (CVD) are a group of illnesses that include coronary heart disease, cerebrovascular disease, congenital heart disease, and deep vein thrombosis. CVD is the leading cause of mortality worldwide, representing 31% of deaths. In Spain, CVD caused 24% of all deaths in 2020. Major surgery is often chosen as the treatment of choice for CVD. The concept of fast-track rehabilitation after surgery appeared in the 1970s. Participation in these exercise-based prehabilitation programs may decrease postoperative complications and length of hospital stay.

The purpose of the present study is to evaluate whether the implementation of an additional resistance training (RT) prehabilitation protocol within a cardiac exercise-based prehabilitation can reduce ICU length of stay, postoperative complications, and hospital length of stay (LOS). Additionally, the secondary objective is to determine whether a program that includes RT in addition to respiratory and aerobic training can have better effects on ventilatory variables.

This study follows the protocol of a prospective, parallel, non-randomized clinical trial. Ninety-six adult patients diagnosed with valvular pathology and who have been scheduled for surgery will be included. The control group will be treated with ventilatory and strengthening of respiratory muscles, as well as aerobic exercise. The experimental group, in addition, will receive RT targeting peripheral muscles. Variables such as hospital stay, quality of life, respiratory values, and exercise capacity will be evaluated. Quantitative variables will be analyzed using a t-test or ANOVA, or Mann-Whitney test if the distribution is non-parametric.

ELIGIBILITY:
Inclusion Criteria:

* adult patients diagnosed with valvular pathology who have been admitted as candidates for cardiac surgery for the first time, and who have been scheduled for surgery

Exclusion Criteria:

* stage 4 or 5 renal failure, low ejection fraction, Euroscore greater than 15 (Nashef et al., 2012) , non-ST-segment elevation acute coronary syndrome (NSTEACS), coronary artery disease, or need for urgent intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
length of stay in hospital | 1 year
  length of hospital stay from admission to discharge
Length of stay in ICU | 1 year
  length of ICU stay from admission until the transfer of the patient to his room
EuroQoL-5D | 1 year
  Perception of quality of life

SECONDARY OUTCOMES:
Inspiratory capacity | 1 year
  the volume of air that can be inspired by the resting inspiratory position
Peak expiratory flow | 1 year
  the maximum flow that a person can exhale during a brief maximal expiratory effort after full inspiration
Respiratory pressures | 1 year
  the strength of the respiratory muscles, both at diaphragmatic (inspiratory) and abdominal and intercostal (expiratory) levels
Exercise capacity | 1 year
  Patient's ability to perform physical exertion

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de La Ribera, Alzira, Alzira, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided